CLINICAL TRIAL: NCT04398199
Title: A Single Arm Phase II Study of Hypofractionated Radiotherapy Alone in Locally Advanced Nonsmall Cell Lung Cancer Patients Who Decline or Are Ineligible for Surgery or Chemotherapy
Brief Title: Study of Hypofractionated Radiotherapy Alone in Locally Advanced Nonsmall Cell Lung Cancer Patients
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Low accruals
Sponsor: Wake Forest University Health Sciences (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IRB00065905; WFBCCC 62220 (Other: Wake Forest Baptist Comprehensive Cancer Center)
Record Dates: First submitted 2020-05-18; First posted 2020-05-21 (Actual); Results first posted 2022-10-05 (Actual); Last update posted 2022-10-05 (Actual); Status verified 2022-09

CONDITIONS: Nonsmall Cell Lung Cancer, Stage II; Nonsmall Cell Lung Cancer Stage III
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Hypofractionated Radiation Therapy (Experimental): Hypofractionated radiation therapy will be delivered to all participants. The radiation will be planned in a special way to give the biggest parts of the tumors that are the most difficult to control a little more radiation every day than the lower risk areas.
  Interventions: Drug: Hypofractionated Radiation Therapy; Radiation: Radiation Boost

INTERVENTIONS:
Drug: Hypofractionated Radiation Therapy — The prescribed dose will be 70 Gy in 25 fractions. Participants will radiation therapy once a day for 25 days, Monday through Friday (around 5 weeks).
Radiation: Radiation Boost — Undergo simultaneous integrated boost (SIB) to treat both planned target volumes with daily image guidance. This approach allows daily confirmation of target localization and simultaneous delivery of lower dose per fraction to low risk areas while maintaining a high dose per fraction to the highest risk areas.

SUMMARY:
The purpose of this research study is to find out what effects (good or bad) may come from a new way of doing radiation therapy for lung cancer. This study is for patients who are not able to get surgery or chemotherapy with their radiation. The way of doing radiation therapy in this trial is called hypofractionated radiation therapy which is a standard approach, but this study allows the actual tumor to get an extra radiation dose while still protecting the organs that are near the tumor.

DETAILED DESCRIPTION:
Primary Objective:

• To determine the in-field control of hypofractionated radiotherapy consisting of 70 Gy in 25 fractions without concurrent chemotherapy measured at two years after the first post- radiotherapy scan.

Secondary Objective(s):

* To determine the toxicity profile of thoracic hypofractionated radiotherapy consisting of 70 Gy in 25 fractions as graded by Common Terminology Criteria for Adverse Events (CTCAE) version 5.0
* To determine proportion with local, regional, and distant progression at 1 and 2 years after the first post-radiotherapy scan, and compute progression-free and overall survival (progression-free survival and overall survival, respectively).

ELIGIBILITY:
Inclusion Criteria:

* Histological confirmation of non-small cell lung cancer by either biopsy or cytology
* American Joint Committee on Cancer (AJCC) 8th Edition Stage II-III or ultracentral Stage IB disease as determined by PET/CT and MRI Brain
* Ultracentral disease will be defined as edge of gross visible tumor within 1.0 cm of the proximal bronchial tree.
* Eastern Cooperative Oncology Group (ECOG) Performance Status of 0-3
* Participant is not eligible for or has declined surgical resection or stereotactic body radiotherapy as determined by the treating physician
* Participant is not eligible for or has declined concurrent chemotherapy as determined by the treating physician
* While investigators expect it to be an uncommon event, sequential use of systemic therapy after completion of radiation therapy is permissible if the participant's status improves such that they become eligible for such therapies, per the discretion of a multidisciplinary tumor board.
* Negative serum or urine pregnancy test within 2 weeks of the date of enrollment for women of child-bearing potential.
* Ability to understand and the willingness to sign an IRB-approved informed consent document (either directly or via a legally authorized representative).

Exclusion Criteria:

* History of previous thoracic radiotherapy with the exception of prior radiotherapy for breast cancer without overlap of the fields with the cancer to be treated.
* Prior systemic therapy or surgery for the study cancer.
* Prior malignancy within the past two years except for non-melanoma skin cancer, prostate cancer, or any in-situ malignancy.
* Receipt of anti-angiogenic therapy, such as bevacizumab, within 6 months of enrollment.
* Pregnant women are excluded from this study because radiation therapy has known potential for teratogenic or abortifacient effects.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1 (Actual)
Dates: Start 2020-10-16 (Actual); Primary Completion 2020-11-20 (Actual); Study Completion 2020-11-20 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Michael Farris, MD, Principal Investigator — Wake Forest University Health Sciences
Locations (1):
- Wake Forest Baptist Comprehensive Cancer Center, Winston-Salem, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Hypofractionated Radiation Therapy
Started | 1
Completed | 1
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Hypofractionated Radiation Therapy
Number analyzed (Participants) | 1
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 1
  >=65 years | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 1
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 1
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 1
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 1

OUTCOME MEASURES:

1. Primary Outcome: Presence or Absence of In-Field Progression
Description: In-field progression is defined as growth of the targeted lesions beyond the treated volume. The treated volume will be defined as the 28.75 Gy isodose line (50% of 57.5 Gy). Pathologic confirmation of tumor progression is preferred, but can be determined radiographically by Multidisciplinary Thoracic Oncology Program consensus if biopsy of the lesion in question is not feasible or safe. Investigators will compare the proportion of the sample with any in-field progression at 2 years to the historical control proportion of 0.5, using a one-sample z-test.
Time Frame: At 2 years
Population: Study was terminated early due to low accruals, outcome measure data not available.
Arm/Group | Hypofractionated Radiation Therapy
Number analyzed (Participants) | 0

2. Secondary Outcome: Proportion of Participants Experiencing Grade 2 or Higher Toxicities
Description: Toxicities will be evaluated per Common Terminology Criteria for Adverse Events (CTCAE) Version 5.0 constructed with a 95% confidence interval.
Time Frame: 25 months
Population: Study was terminated early due to low accruals, outcome measure data not available.
Arm/Group | Hypofractionated Radiation Therapy
Number analyzed (Participants) | 0

3. Secondary Outcome: Proportion of Participants That Experienced Local Progression
Description: Participants who have experienced local progression by 13 months (1 year following first post-radiotherapy scan) and by 25 months (2 years following first post-radiotherapy scan), and will also compute the same two proportions considering regional progression, distant progression, and any (of the 3 categories) progression. A 95% confidence intervals around these proportions will be constructed. Participants for whom investigators are unable to determine progression status at 1 and 2 years (e.g., because they do not return for the necessary scans, or because they die without evidence of progression) will be left out of these analyses.
Time Frame: At 1 and 2 years after first post-radiotherapy scan
Population: Study was terminated early due to low accruals, outcome measure data not available.
Arm/Group | Hypofractionated Radiation Therapy
Number analyzed (Participants) | 0

4. Secondary Outcome: Progression-Free Survival
Description: Progression-free survival will be evaluated by considering the time from registration to progression of disease or death; those who do not experience either outcome will be censored at date of last visit. Using the Kaplan-Meier lifetable method, and will estimate median survival and corresponding 95% confidence intervals; investigators will also explore simple Cox proportional hazards models of this survival outcomes, to examine the predictive influence of variables such as age, gender, ECOG performance status, stage at diagnosis, planning target volume (PTV) 7000 volume, and planning target volume (PTV) 5750 volume.
Time Frame: Up to 2 years
Population: Study was terminated early due to low accruals, outcome measure data not available.
Arm/Group | Hypofractionated Radiation Therapy
Number analyzed (Participants) | 0

5. Secondary Outcome: Overall Survival
Description: Overall survival will be evaluated by considering the time from registration to death from any cause; those who do not die will be censored at date of last visit. Using the Kaplan-Meier lifetable method, and will estimate median survival and corresponding 95% confidence intervals; investigators will also explore simple Cox proportional hazards models of this survival outcomes, to examine the predictive influence of variables such as age, gender, ECOG performance status, stage at diagnosis, planning target volume (PTV) 7000 volume, and planning target volume (PTV) 5750 volume.
Time Frame: Up to 2 years
Population: Study was terminated early due to low accruals, outcome measure data not available.
Arm/Group | Hypofractionated Radiation Therapy
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Time Frame: Up to 3 months
Arm/Group | Hypofractionated Radiation Therapy
All-Cause Mortality (participants affected / at risk) | 1/1
Serious Adverse Events (participants affected / at risk) | 1/1
Other Adverse Events (participants affected / at risk) | 1/1
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Hypofractionated Radiation Therapy (N=1)
Acute kidney injury (Renal and urinary disorders) | 1 (1)
Hyperglycemia (Metabolism and nutrition disorders) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Hypofractionated Radiation Therapy (N=1)
Skin ulceration (Skin and subcutaneous tissue disorders) | 1 (1) — Pressure ulcer
Constipation (Gastrointestinal disorders) | 1 (1)
Fever (General disorders) | 1 (1)
Sepsis (Infections and infestations) | 1 (1)
Hip fracture (Injury, poisoning and procedural complications) | 1 (1)
Fatigue (General disorders) | 1 (1)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Gastrointestinal disorder, other (Gastrointestinal disorders) | 1 (1) — Thrush
Blood and lymphatic disorders, other (Blood and lymphatic system disorders) | 1 (1) — Thrombolic event

LIMITATIONS AND CAVEATS:
One patient was accrued to this trial. He was assigned to the intervention arm. He began on study on 10/16/2020, and began treatment on 10/19/2020. He went off treatment 11/20/2020 due to a fall-he did not return for follow-up after week 3. He expired on 1/8/2021. The study was terminated early due to slow accruals which did not allow enough time for data collection for any outcome measures to properly assess the clinical trial.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2021-04-22): https://cdn.clinicaltrials.gov/large-docs/99/NCT04398199/Prot_SAP_001.pdf
  • Informed Consent Form (2021-05-24): https://cdn.clinicaltrials.gov/large-docs/99/NCT04398199/ICF_000.pdf